CLINICAL TRIAL: NCT05909631
Title: Comparing Effects of Beetroot Juice and Mediterranean Diet on Liver Enzymes and Sonography in Patients With Non-Alcoholic Fatty Liver Disease (NAFLD): A Randomized Control Trials
Brief Title: Comparing Effects of Beetroot Juice and Mediterranean Diet on Liver Enzymes and Sonography in Patients With NAFLD
Acronym: BJ
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sulaimany Polytechnic university (Other)
Responsible Party: Principal Investigator, Hawal Lateef Fateh, Dr Hawal Lateef Fateh, Sulaimany Polytechnic university
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KTC1212
Record Dates: First submitted 2023-05-10; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: NAFLD, Non-alcoholic Fatty Liver Disease
Keywords: Mediterranean diet; Beetroot juice; nonalcoholic fatty liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Diet, Mediterranean

STUDY DESIGN:
Intervention Model Description: The participants were split into four groups: control, Mediterranean diet with beet juice (BJ+MeD), Mediterranean diet alone (MeD) and beetroot juice (BJ). The Mediterranean diet included fruits, vegetables, fish, poultry, and other lean meats (without skin), sources of omega-3 fatty acids, nuts, and legumes. Beetroot juice had 250 mg of beetroot.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Statical analyser
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- 250 ml of a placebo (Placebo Comparator): 250 ml of a placebo
  Interventions: Other: placebo
- beetroot juice (BJ) (Experimental): 250 ml of concentrated beetroot juice
  Interventions: Other: Beetroot juice
- Mediterranean diet with beet juice (BJ+MeD) (Experimental): Mediterranean diet with beet juice (BJ+MeD)
  Interventions: Combination Product: Mediterranean diet with beet juice (BJ+MeD)
- Mediterranean diet alone (MeD) (Experimental): Mediterranean diet alone (MeD)
  Interventions: Other: Mediterranean diet alone (MeD)

INTERVENTIONS:
Other: Beetroot juice — 250 ml of concentrated beetroot juice, were given to participants in the BJ groups .This was carried out in the morning, 30 minutes before breakfast, and on an empty stomach.
  Arms: beetroot juice (BJ)
Other: placebo — 250 ml of a placebo
  Arms: 250 ml of a placebo
Other: Mediterranean diet alone (MeD) — Mediterranean diet alone (MeD)
  Arms: Mediterranean diet alone (MeD)
Combination Product: Mediterranean diet with beet juice (BJ+MeD) — Mediterranean diet with beet juice (BJ+MeD).
  Arms: Mediterranean diet with beet juice (BJ+MeD)

SUMMARY:
The goal of this clinical trial study is to investigate comparing Effects of Beetroot juice and Mediterranean diet on Liver Enzymes and Sonographic appearance in Patients with Non-Alcoholic Fatty Liver Disease (NAFLD)

The main question[s] it aims to answer are:

1. Beetroot juice has role in reduce Liver Enzymes
2. Mediterranean diet has role in reduce Liver Enzymes

DETAILED DESCRIPTION:
Patients with NAFLD were identified and enrolled for this research at the PAR hospital in the Kurdistan Region of Iraq.

For 12 weeks, for the group members who were receiving the MeD, we recommended consuming Mediterranean foods like fish, poultry, sources of omega-3, vegetables and colored fruits, legumes and nuts, and low-fat goods while avoiding inflammatory foods like high-fat foods, processed meats, fast food, simple sugars, chips, and soft drinks.

At baseline, the participants' demographic and anthropometric information, including as gender, age, weight, height, smoking status, location of residence, and physical activity, were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients had to be between the ages of 19 and 73, and they had to have NAFLD as their main diagnosis.
2. For a NAFLD diagnosis, ultrasound proof of fatty liver (stage I or above) and an elevated level of liver enzymes were required.

Exclusion Criteria:

1. history of diseases like cardiovascular, liver, chronic hepatitis C, and kidney disease
2. supplement use within the previous six months; hormone therapy; use of drugs like amiodarone, methotrexate, and corticosteroids
3. cases of starvation or inadequate nutrition; pregnancy; metabolic disorders like Wilson disease and glycogen storage disease; a history of liver irradiation

Ages: 19 Years to 73 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-04-11 (Actual)

PRIMARY OUTCOMES:
Beetroot juice has role in reduce liver enzymes | 12 weeks
  Beetroot juice was given for 12 weeks and has role in reduce Serum Bilirubin, alkaline phosphatase (ALP), alanine transaminase (ALT), and liver enzyme was measured by blood sampling tests.

SECONDARY OUTCOMES:
Mediterranean diet contributes to lower liver enzyme levels. | 12 weeks
  Mediterranean diet was given for 12 weeks and has role in reduce Serum Bilirubin, alkaline phosphatase (ALP), alanine transaminase (ALT), and liver enzyme was measured by blood sampling tests.

CONTACTS AND LOCATIONS:
Overall Officials: Hawal Lateef, Msc, Principal Investigator — Nursing department, sulaimany polytechni university, kurdistan, iraq
Locations (1):
- Hawal, Sulaymaniyah, Sulaimanyah, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fateh HL, Rashid SA, Muhammad SS, Al-Jaf SH, Ali AM. Comparing effects of beetroot juice and Mediterranean diet on liver enzymes and sonographic appearance in patients with non-alcoholic fatty liver disease: a randomized control trials. Front Nutr. 2023 Aug 17;10:1181706. doi: 10.3389/fnut.2023.1181706. eCollection 2023. PMID 37662597